CLINICAL TRIAL: NCT05526417
Title: Pre-Operative ERAS® (Enhanced Recovery After Surgery): Randomized Feasibility Trial of Implementing Individualized Prehabilitation for People Undergoing Neo-Adjuvant Radiotherapy and Lower Limb Soft-Tissue Sarcoma Surgery
Brief Title: Individualized Prehabilitation for Enhancing Recovery and Surgical Outcomes in Patients Undergoing Radiotherapy and Surgery for Soft Tissue Sarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GMROA2182; NCI-2022-05583 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-002674 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Sarcoma; Stage I Soft Tissue Sarcoma of the Trunk and Extremities; Stage II Soft Tissue Sarcoma of the Trunk and Extremities; Stage III Soft Tissue Sarcoma of the Trunk and Extremities
MeSH Terms: conditions — Sarcoma | interventions — Early Intervention, Educational; Educational Status; Methods; Magnetic Resonance Spectroscopy; Physical Therapy Modalities; Telemedicine

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Masking of treatment assignment to the surgeon and radiation oncologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (prehabilitation physical therapy) (Experimental): Patients perform personalized prehabilitation physical therapy exercises BID 5 days per week for 8 weeks while receiving standard of care radiotherapy and prior to standard of care surgery, attend telemedicine visits with a physical therapist once a week for 9 weeks, and receive educational materials. Patients undergo MRI and CT at week 9.
  Interventions: Procedure: Computed Tomography; Other: Educational Intervention; Procedure: Magnetic Resonance Imaging; Procedure: Physical Therapy; Other: Questionnaire Administration; Other: Telemedicine
- Arm II (educational materials) (Active Comparator): Patients receive educational materials and attend a telemedicine visit with a research assistant once a week for 8 weeks while receiving standard of care radiotherapy and prior to standard of care surgery. Patients undergo MRI and CT at week 9.
  Interventions: Procedure: Computed Tomography; Other: Educational Intervention; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Other: Telemedicine

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Educational Intervention — Receive educational materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Physical Therapy — Receive prehabilitation physical therapy
  Other Names: Physiatric Procedure; Physical Medicine Procedure; Physical Therapeutics; Physical Therapy Procedure; Physiotherapy; Physiotherapy Procedure; PT
  Arms: Arm I (prehabilitation physical therapy)
Other: Questionnaire Administration — Ancillary studies
Other: Telemedicine — Attend telemedicine visits
  Other Names: Telehealth

SUMMARY:
This clinical trial evaluates whether patients with deep soft tissue sarcomas who receive a tailored prehabilitation exercise regimen during standard radiotherapy and prior to standard of care surgery have better recovery and surgical outcomes than those who do not. Patients undergoing surgery to soft tissue sarcomas are at high risk for post-operative disability, which is associated with high rates of depression and poor health-related quality of life. Prehabilitation is the practice of exercising before surgery to ensure that the patient is in the best possible condition. It allows patients to prepare their bodies for recovery after surgery, which may result in better surgical outcomes, recovery, and quality of life after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if a tailored prehabilitation program focusing on functional optimization of spared limb tissue in two groups of patients with localized, lower extremity soft tissue sarcoma, one with prehabilitation and one with equal attention and informational support, improves functional outcome as measure by the Toronto Extremity Salvage Score (TESS).

II. To identify the measures and metrics most responsive to the intervention using the (TESS), Six Minute Walk Test (6MWT), wearable Heel2Toe sensor technology, and daily step count.

III. To estimate recruitment, retention, adherence, and acceptability rates.

SECONDARY OBJECTIVES:

I. To compare changes in quality of life over time as a result of the prehabilitation intervention using the Edmonton Symptom Assessment Scale (ESAS), European Quality of Life Five Dimension Five Level Scale Questionnaire (EQ-5D-5L) (Euroqol Group), the Patient Generated Index (PGI).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients perform personalized prehabilitation physical therapy exercises twice a day (BID) 5 days per week for 8 weeks while receiving standard of care radiotherapy and prior to standard of care surgery, attend telemedicine visits with a physical therapist once a week for 9 weeks, and receive educational materials. Patients undergo magnetic resonance imaging (MRI) and computed tomography (CT) at week 9.

ARM II: Patients receive educational materials and attend a telemedicine visit with a research assistant once a week for 8 weeks while receiving standard of care radiotherapy prior to standard of care surgery. Patients undergo MRI and CT at week 9.

After completion of study, patients are followed up at weeks 2, 6, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-proven deep soft tissue sarcoma (STS) of the lower extremity
* Localized
* Adults, 18 and older
* All gender types
* Subjects must be able to provide appropriate consent or have an appropriate representative available to do so

Exclusion Criteria:

* Soft tissue sarcomas that are in a superficial location relative to fascia
* Patients with metastatic disease (distant or nodal)
* Both and upper and lower extremity involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by recruitment, retention, adherence, and acceptability | Up to 22 weeks
  Univariate descriptive statistics and frequency distributions will be calculated, as appropriate for all variables. Baseline values for demographic, clinical, and outcome variables will be tabulated for the treatment groups.
Efficacy potential | Up to 22 weeks
  Univariate descriptive statistics and frequency distributions will be calculated, as appropriate for all variables. Baseline values for demographic, clinical, and outcome variables will be tabulated for the treatment groups. Between-group effect sizes will be estimated for continuous outcomes.
Toronto Extremity Salvage Score | At 2, 6, and 12 weeks
  This is a self-report measure comprising 30 items (23 for activities of daily living; 7 items for role participation). Will use this measure, completed using observed performance for feasible items and self-report for the remaining items (getting in and out of a car, shopping; driving). Univariate descriptive statistics and frequency distributions will be calculated, as appropriate for all variables. Baseline values for demographic, clinical, and outcome variables will be tabulated for the treatment groups. Between-group effect sizes will be estimated from a mixed model which considers the individual as a cluster with multiple measures per person.
Functional walking capacity | At 2, 6, and 12 weeks
  Functional walking capacity is defined as walking capacity needed for everyday activities of daily living such as shopping, traveling to and from work, and walking in the workplace or public buildings. The six minute walk test (6MWT) is the gold standard measure for this. The units are distance in meters covered during the test. There is a standardized mobile application for measuring and data comes minute by minute to assess fatigability. Univariate descriptive statistics and frequency distributions will be calculated, as appropriate for all variables.
Gait quality | Up to 22 weeks
  Gait quality will be measured during the 6MWT using a wearable developed by the team, Heel2Toe sensor. The parameters of gait quality will include proportion of steps with as strong a heel strike pre-operatively, as well as distribution of cadence and of angular velocity. Irregular stepping pattern is indicated by lack of heel strike, large variability in cadence, stride length, and angular velocity as indicated by coefficient of variation. Univariate descriptive statistics and frequency distributions will be calculated, as appropriate for all variables.
Daily step count | Up to 22 weeks
  Daily step count for the duration of the study will be obtained using the native accelerometer/gyroscope and pedometers available on both iPhone and android devices. Will summarize this complex data using benchmarks of 1, 3, 5, 7, 9 (000 steps) based on meaningful physical activity targets. Will measure the time to achieve these targets post-surgery. These will be captured for the 9 week prehabilitation period and the post-surgery recovery period. As indicated, will focus on steps taken outside of the house as "in house" steps tend to be of very low cadence. For step counts, time to reach the benchmarks of 1, 3, 5, 7, 9 (000 steps) will be calculated and presented descriptively. Univariate descriptive statistics and frequency distributions will be calculated, as appropriate for all variables.

SECONDARY OUTCOMES:
Symptom status | Up to 22 weeks
  Symptom status will be assessed using the Edmonton Symptom Assessment Scale which assesses 7 symptoms including pain, fatigue, distress, and overall well-being. Univariate descriptive statistics and frequency distributions will be calculated, as appropriate for all variables.
Global health related quality of life | Up to 22 weeks
  Global health related quality of life will be measured using the 5-level EQ-5D version (Euroqol Group) and the Patient Generated Index will be used to assess quality of life. Univariate descriptive statistics and frequency distributions will be calculated, as appropriate for all variables.

CONTACTS AND LOCATIONS:
Overall Officials: Krista A. Goulding, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials